CLINICAL TRIAL: NCT03303469
Title: Hypoxic Changes in Hepatocellular Carcinoma (HCC) Following Trans Arterial Chemo Embolization and Stereotactic Radiation: [18F]Fluoromisonidazole (FMISO) Imaging
Brief Title: Hypoxic Changes in Hepatocellular Carcinoma (HCC) Following Trans Arterial Chemo Embolization and Stereotactic Radiation: Fluorine18 (18F) Fluoromisonidazole (FMISO) Imaging
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study was terminated due to poor enrollment
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Janis P. O'Malley, MD, Principal Investigator, Professor of Radiology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: F170519002
Record Dates: First submitted 2017-09-13; First posted 2017-10-06 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — fluoromisonidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FMISO PET imaging post TACE and Stereotactic body radiation therapy (SBRT) (Experimental): FMISO imaging at baseline, post-TACE and post-SBRT
  Interventions: Drug: FMISO

INTERVENTIONS:
Drug: FMISO — FMISO PET/CT imaging at baseline
Drug: FMISO — FMISO PET/CT post TACE
Drug: FMISO — FMISO PET/CT post SBRT

SUMMARY:
[18F] FMISO Positron Emission Tomography (PET) to determine hypoxia in patients with HCC treated with TACE.

DETAILED DESCRIPTION:
This Phase II study will investigate the utility of [18F] FMISO in patients with hepatocellular carcinoma (HCC). This trial is designed to test the hypothesis that PET determined [18F]FMISO uptake will indicate tumor hypoxia in patients with HCC treated with trans-arterial chemo-embolization (TACE). We anticipate that [18F] FMISO PET/CT will advance our understanding of the role of hypoxia in HCC prior to treatment and that this knowledge will help design newer combination therapeutic trials for better treatment outcomes. [18F] FMISO PET/CT provides three parameters, tissue hypoxic volume (HV), maximum tissue to blood uptake ratio (T:Bmax) and tumor blood flow. Both pre-and post-therapy images will be examined to investigate changes in these parameters during the course of TACE treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years of age) patients with documented HCC tumor mass >3cm, who are scheduled to undergo TACE with additional selective internal radiation therapy (SIRT)
* The appropriate criteria for inclusion for this patient population are:
* Biopsy or radiological diagnosis of HCC (defined as Organ Procurement and Transplantation Network (OPTN*) Category 5 lesion either on CT or MRI)
* Scheduled for TACE (using doxorubicin-eluting beads) + SBRT
* Willingness to undergo PET/CT
* Able to lie on the imaging table for up to 1 hour.
* Able to provide signed informed consent.
* Women with childbearing potential must have a negative urine Beta-Human Chorionic Gonadotropin (β-hCG) test day of procedure

Exclusion Criteria:

* Estimated life expectancy <12 months or serious medical co-morbidities that would preclude definitive local therapy
* Unable to lie on the imaging table
* Age less than 18 years.
* Pregnancy or lactation
* Inability or unwillingness to provide informed consent.
* Weight >500 lbs (the weight limit of the tomograph gantry table)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janis P O'Malley, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Advanced Imaging Facility, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FMISO PET Imaging Post TACE and SBRT: FMISO imaging at baseline, post-TACE and post-SBRT
  FMISO: FMISO PET/CT imaging at baseline
  FMISO: FMISO PET/CT post TACE
  FMISO: FMISO PET/CT post SBRT
Period: Overall Study
Arm/Group | FMISO PET Imaging Post TACE and SBRT
Started | 3
Completed | 1
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | FMISO PET Imaging Post TACE and SBRT
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Quantitate HCC Tumor Hypoxia at Baseline Using FMISO Positron Emission Tomography (PET).
Description: Perform PET/CT imaging using FMISO at baseline to measure tumor hypoxia
Time Frame: At baseline
Population: We were unable to perform the statistical analysis due to insufficient data collection.
Arm/Group | FMISO PET Imaging Post TACE and SBRT
Number analyzed (Participants) | 0

2. Primary Outcome: Measure Changes in HCC Tumor Hypoxia and Blood Flow After Trans-arterial Chemoembolization (TACE), Prior to Radiotherapy.
Description: Perform PET/CT imaging using FMISO post-TACE and prior to Stereotactic body radiation therapy (SBRT) to determine tumor hypoxia
Time Frame: 1 month post-TACE procedures and prior to SBRT
Population: We were unable to perform the statistical analysis due to insufficient data collection.
Arm/Group | FMISO PET Imaging Post TACE and SBRT
Number analyzed (Participants) | 0

3. Primary Outcome: Measure Changes in Treated HCC Tumor Hypoxia Following TACE and Radiotherapy
Description: Perform PET/CT imaging using FMISO post-SBRT to determine tumor hypoxia
Time Frame: 1 month post-SBRT
Population: We were unable to perform the statistical analysis due to insufficient data collection.
Arm/Group | FMISO PET Imaging Post TACE and SBRT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Between 4 to 6 weeks.
Arm/Group | FMISO PET Imaging Post TACE and SBRT
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT03303469/Prot_SAP_001.pdf